CLINICAL TRIAL: NCT04342104
Title: NIV and CPAP Failure Predictors in COVID-19 Associated Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Morales Meseguer (Other)
Responsible Party: Principal Investigator, Miguel Filipe Martins de Matos Navarro Guia, Dr., Hospital General Universitario Morales Meseguer
Other Study IDs: 08-04-2020
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Failure; Covid-19
Keywords: noninvasive ventilation; CPAP; Covid-19; Respiratory failure; HACOR score
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for biochemistry and blood count
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NIV: Patients on Bilevel NIV
  Interventions: Other: Monitoring for aggravation; Other: Evaluate HACOR score effectivity in this patients
- CPAP: Patients on CPAP
  Interventions: Other: Monitoring for aggravation; Other: Evaluate HACOR score effectivity in this patients

INTERVENTIONS:
Other: Monitoring for aggravation — Monitor patients on CPAP or NIV and analyzing possible variables that may predict failure, namely:
  * lymphopenia
  * thrombocytopenia
  * CRP
  * ferritin
  * LDH
  * troponin I
  * NT-ProBNP
  * Liver enzymes
  * D-dimers
  * radiologic aggravation " 1 day and 1 week after starting NIV or CPAP
Other: Evaluate HACOR score effectivity in this patients — Apply the HACOR score after starting NIV and CPAP and later verify if it was effective in predicting NIV/CPAP failure

SUMMARY:
Evaluate HACOR socre utility and efficacy in predicting NIV and/or CPAP failure in patients with COVID-19 associated respiratory failure.

Propose adaptations to HACOR score based on the "state of art" of COVID-19

DETAILED DESCRIPTION:
Evaluate HACOR socre utility and efficacy in predicting NIV and/or CPAP failure in patients with COVID-19 associated respiratory failure.

Propose adaptations to HACOR score based on the "state of art" of COVID-19

- this adaptations may include radiologic aggravation and monitoring of CRF, ferritin, LDH, d-dimers, NT-proBNP, troponin I, GOT, GPT, blood count

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute respiratory failure due to COVID-19 who have initiated NIV or CPAP based on assistant clinician decision

Exclusion Criteria:

* Patients with imediate indication to invasive mechanical ventilation
* Patients with any formal contraindication to noninvasive respiratory support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory failure due to COVID-19 who have initiated NIV or CPAP based on assistant clinician decision
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
HACOR score efficacy | 1 hour after initation of CPAP or NIV
  Analyze if HACOR score is effective in predicting nonivasive ventilation failure in COVID-19 associated respiratory failure
HACOR score addaptation | 1 - 2 weeks
  Analyze the role of possible variables to be added to HACOR score in order to improve efficay in COVID-19 patients

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Guia, Principal Investigator — Hospital General Universitario Morales Meseguer; Antonio Esquinas, Study Director — Hospital General Universitario Morales Meseguer
Locations (1):
- Hospital General Universitario Morales Meseguer, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided